CLINICAL TRIAL: NCT03053947
Title: Pain Free Laceration Repairs Using Intra-nasal Ketamine: A Dose Escalation Clinical Trial
Brief Title: Pain Free Laceration Repairs Using Intra-nasal Ketamine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Evelyne D.Trottier (Other)
Responsible Party: Sponsor-Investigator, Evelyne D.Trottier, M.D., FRCPC, St. Justine's Hospital
Organization: St. Justine's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-1149
Record Dates: First submitted 2016-12-22; First posted 2017-02-15 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Laceration
Keywords: Intranasal Ketamine; Pain Management
MeSH Terms: conditions — Lacerations; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ketamine IN (Other): All participants will receive intranasal Ketamine between 3mg/kg up to 9 mg/kg, once.
  Interventions: Drug: Intranasal Ketamine

INTERVENTIONS:
Drug: Intranasal Ketamine — Administration of intranasal ketamine at a dose from 3 to 9 mg/kg for safe and effective procedural sedation for laceration repair in the ED for children aged 1 to 12 year-old.

SUMMARY:
Lacerations are one of most common trauma in children presenting to the emergency department (ED). Currently, there are wide variations regarding sedation and analgesia practices when suture are required. Even though topical anesthesia is very useful to reduce pain, it does not obviate the use of pharmacologic agents to decrease stress in anxious children undergoing laceration repairs in the ED.

There is a growing interest in the intranasal (IN) route of administration in the pediatric population. It bypasses the first hepatic passage and thus provides medications direct access to the systemic circulation leading to higher and faster serum concentrations than would the oral route. Also, intravenous (IV) cannulation can be avoided reducing the pain associated with it and the need for nursing time and procedure delay. IN fentanyl and midazolam are two agents that can be combined for this procedure, but respiratory depression is a feared adverse effects. Ketamine is the most commonly used IV agent for procedural sedation, and can offer potent analgesia and sedation while maintaining respiratory drive and protective airway reflexes. Few studies have evaluated IN ketamine for procedural sedation. There is a wide range of dosing reported from 3 to 9 mg/kg. This raises the question as what is the lowest possible dosage that can be used to successfully repairs laceration in children with minimal restrain and no adverse events, as described by the Pediatric Emergency Research Canada (PERC)/ Pediatric Emergency Care Applied Research Network (PECARN) consensus.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 1 to 12 years;
2. Weight between 10 and 30 kg
3. Any laceration requiring sutures repair;
4. Need for procedural sedation according to the emergency physician assessment for the suture repair

Exclusion Criteria:

1. American Society of Anesthesiologists (ASA) physical status class III and more;
2. Previous administration of IV, IN or oral analgesics or opioid other than acetaminophen and ibuprofen;
3. Allergy or previous adverse reaction to ketamine;
4. Aberrant nasal anatomy or nasal trauma;
5. Presence of multiple trauma or eye rupture suspicion
6. Head injury with loss of consciousness, decreased Glasgow Coma Scale (GCS) or intracranial bleeding;
7. Cognitive impairment;
8. Known glaucoma;
9. Pregnancy
10. Language barrier
11. Known schizophrenia or psychotic event;
12. Uncontrolled hypertension;
13. Airway instability (tracheal surgery, tracheal stenosis, tracheomalacia, and laryngomalacia)
14. Active pulmonary infections (including upper respiratory infections)
15. Known or suspected cardiac disease
16. Known or suspected kidney disease

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2019-11-27 (Actual)

PRIMARY OUTCOMES:
DosINK 1-Optimal dose of intranasal ketamine for adequate procedural sedation as assessed by the PERC/PECARN consensus criteria for procedural sedation in children during their laceration repair. | 18 months
  Dose finding : determine the optimal dose of IN ketamine between a range of 3 and 9 mg/kg for laceration suture repair
DosINK 2- Evaluation of the dose determined in DosINK 1 of intranasal ketamine for adequate procedural sedation as assessed by the PERC/PECARN consensus criteria for procedural sedation in children during their laceration repair. | 18 months
  Dose evaluation: Evaluate the dose determined in DosINK 1 in 30 patients

SECONDARY OUTCOMES:
Pain before, during and after the procedure assessed with the Faces pain scale Revised for children older than 4 year-old and with the Face Legs Activity Cry Consolability (FLACC) score for children younger than 4 year-old. | 18 months
Anxiety before, during and after the procedure assessed with the Procedure behavioural rating revised scale. | 18 months
Sedation level during the procedure and time to return to baseline using the University of Michigan sedation scale (UMSS). | 18 months
Parents, patients and provider satisfaction with sedation as assessed by Likert scale. | 18 months
Sides effects and adverse events as assessed by the PERC/PECARN consensus criteria for procedural sedation in children. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Evelyne D Trottier, MD, FRCPC, Principal Investigator — St. Justine's Hospital
Locations (2):
- Canada (2):
  - Sickkids, Toronto, Ontario
  - St. Justine's Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rached-d'Astous S, Finkelstein Y, Bailey B, Marquis C, Lebel D, Desjardins MP, Trottier ED. Intranasal ketamine for procedural sedation in children: An open-label multicenter clinical trial. Am J Emerg Med. 2023 May;67:10-16. doi: 10.1016/j.ajem.2023.01.046. Epub 2023 Jan 30. PMID 36774905
- [Derived] Rached-d'Astous S, Bailey B, Marquis C, Lebel D, Desjardins MP, Trottier ED. Laceration repair using intranasal ketamine: a phase 2 dose escalation clinical trial. CJEM. 2022 Apr;24(3):347-348. doi: 10.1007/s43678-021-00235-3. Epub 2021 Dec 20. No abstract available. PMID 34928491